CLINICAL TRIAL: NCT01987518
Title: French Digestive Polyposis Cohorte
Brief Title: French Digestive Polyposis Cohorte Family Adenomatous Polyposis With APC and MYH Gene Mutations , Cowden's Disease With PTEN Gene Mutation, Peutz Jeghers Disease With STK 11 Gene Mutation ,juvénil Polyposis With SMAD 4 Gene Mutation , Serrated and Hyperplastic Polyposis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Principal Investigator, Hôpital Edouard Herriot
Other Study IDs: Peps Data Base; SISRA (Other: SISRA)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Genetic Diagnostic
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- digestive polyposis: Family adenomatous polyposis (APC or MYH genes) Peutz Jeghers Disease Cowden Disease Festooned Polyposis Juvenile Polyposis Hyperplastic Polyposis
  Interventions: Other: Procedure surgery behavioral and genetic diagnosis; Procedure: quality of life after different type of surgery

INTERVENTIONS:
Other: Procedure surgery behavioral and genetic diagnosis — Observational Study
Procedure: quality of life after different type of surgery

SUMMARY:
French cohorte about polyposis digestive diseases

DETAILED DESCRIPTION:
Family Adenomatous Polyposis APC and MYH Genes Peutz Jeghers Disease Cowden Disease Festooned polyposis Juvenile polyposis Hyperplastic polyposis

ELIGIBILITY:
Inclusion Criteria:

* APC Gene mutation
* MYH Homozygote mutation
* COWDEN Disease with PTEN gene mutation
* Peutz Jeghers Disease with STK 11 gene mutation
* Juvenile polyposis with SMAD 4 gene mutation

Exclusion Criteria:

* heterozygote MYH Gene Mutation

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Digestive Polyposis Cohort
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
genetic diagnosis or over 50 polyps in the stomach in the duodenum or in the colon | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: jean christophe saurin, msd, Principal Investigator — HEH Hospital
Locations (1):
- Hopital Edouard Herriot, Lyon, Auvergne-Rhône-Alpes, France